CLINICAL TRIAL: NCT02705300
Title: A Randomized Investigation of Side Effects to FOLFOXIRI in Combination With Tocotrienol or Placebo as First Line Treatment of Metastatic Colorectal Cancer
Brief Title: Side Effects to FOLFOXIRI + Tocotrienol/Placebo as First Line Treatment of Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FOLFOXIRI-Toco
Record Dates: First submitted 2016-02-26; First posted 2016-03-10 (Estimated); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; Oxaliplatin; Leucovorin; Fluorouracil; Tocotrienols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chemotherapy plus tocotrienol (Experimental): Every 2 weeks: irinotecan 165 mg/m2 iv, oxaliplatin 85 mg/m2 iv, calcium folinate 200 mg/m2 iv, and 5-fluorouracil 3200 mg/m2 as a 46 hour infusion.
  Daily: Tocotrienol 300 mg x 3 daily
  Interventions: Drug: Irinotecan 165 mg/m2 iv; Drug: Oxaliplatin 85 mg/m2 iv; Drug: Calcium folinate 200 mg/m2 iv; Drug: 5-fluorouracil 3200 mg/m2; Dietary Supplement: Tocotrienol
- Chemotherapy plus placebo (Placebo Comparator): Every 2 weeks: irinotecan 165 mg/m2 iv, oxaliplatin 85 mg/m2 iv, calcium folinate 200 mg/m2 iv, and 5-fluorouracil 3200 mg/m2 as a 46 hour infusion.
  Daily: Placebo x 3 daily
  Interventions: Drug: Irinotecan 165 mg/m2 iv; Drug: Oxaliplatin 85 mg/m2 iv; Drug: Calcium folinate 200 mg/m2 iv; Drug: 5-fluorouracil 3200 mg/m2; Drug: Placebo

INTERVENTIONS:
Drug: Irinotecan 165 mg/m2 iv — Max. 4 months
Drug: Oxaliplatin 85 mg/m2 iv — Max. 4 months
Drug: Calcium folinate 200 mg/m2 iv — Max. 6 months
Drug: 5-fluorouracil 3200 mg/m2 — Max. 6 months
Dietary Supplement: Tocotrienol — Max. 2 years or at the discretion of the investigator
  Arms: Chemotherapy plus tocotrienol
Drug: Placebo — Max. 2 years or at the discretion of the investigator
  Arms: Chemotherapy plus placebo

SUMMARY:
Treatment with FOLFOXIRI (5-fluorouracil, oxaliplatin, irinotecan) can be effective, but it has serious side effects, which may require hospitalization.

The purpose of this study is to investigate whether the addition of tocotrienol can reduce the side effects to FOLFOXIRI otherwise leading to hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically verified colorectal adenocarcinoma.
* Patients to receive first line treatment of metastatic disease, including potentially resectable or non-resectable disease
* > 6 months without recurrence after end of adjuvant chemotherapy for radically treated stage II or III colorectal cancer
* Disease evaluable according to RECIST 1.1, but not necessarily measurable disease.
* Age 18-75 years
* Performance status (PS) 0-1. If age 71-75, then PS 0
* Life expectancy > 3 months
* Organ and bone marrow function as follows:

  * Neutrophil count ≥ 1.5 x 10^9/L
  * Thrombocytes ≥ 100 x 10^9/L
  * Total bilirubin ≤ 1.5 x upper level of normal (ULN)
  * Alanine transaminase (ALAT) ≤ 2.5 x ULN (or≤ 5 x ULN in case of liver metastases)
* Fertile women must present negative pregnancy test. Male (with a female fertile partner) as well as female patients must use secure contraceptives during and 6 months after end of treatment.
* Orally and written informed consent to treatment and biobank

Exclusion Criteria:

* Primarily resectable metastases
* Chemotherapy, radiotherapy or immunotherapy within 4 weeks
* Known neuropathy ≥ grade 2
* Serious competitive medical condition
* Other concurrent malignant disease other than non-melanoma skin cancer
* Previous serious and unexpected reactions to 5-fluorouracil, calcium folinate, oxaliplatin, irinotecan or capecitabine.
* Hypersensitivity to one or more of the active substances or auxilliary agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-05-06 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2024-03-27 (Actual)

PRIMARY OUTCOMES:
Time to first serious adverse event | 6 months after the last patient has finished chemotherapy

SECONDARY OUTCOMES:
Number of non-planned hospitalizations calculated from date of first treatment until 1 month after completed chemotherapy | 6 months after the last patient has finished chemotherapy
Duration of non-planned hospitalizations calculated from date of first treatment until 1 month after completed chemotherapy | 6 months after the last patient has finished chemotherapy
Death during treatment calculated from date of first treatment until 1 month after completed chemotherapy | 6 months after the last patient has finished chemotherapy
Response rate | 6 months after the last patient has finished chemotherapy
Progression free survival | 6 months after the last patient has finished chemotherapy
Overall survival | 6 months after the last patient has finished chemotherapy
Number of patients with treatment related adverse events as assessed by CTCAE v.4.0 | 6 months after the last patient has finished chemotherapy
Quality of life as measured by combined questionnaire consisting of EORTC QLQ-C30 and CR29 | 6 months after the last patient has finished chemotherapy
Resection rate | 6 months after the last patient has finished chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Lars H Jensen, PhD, Study Chair — Department of Oncology, Vejle Hospital; Louise R Larsen, MD, Principal Investigator — Department of Oncology, Vejle Hospital
Locations (1):
- Department of Oncology, Vejle Hospital, Vejle, Denmark